CLINICAL TRIAL: NCT02957565
Title: Patient Perception of Physician's Compassion, Communication Skills, and Professionalism During an Outpatient Palliative Care Visit: A Randomized Controlled Trial
Brief Title: Patient Perception of Physician's Compassion, Communication Skills, and Professionalism During an Outpatient Palliative Care Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-0494; NCI-2017-00621 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasms of Independent (Primary) Multiple Sites; Advanced Cancer
Keywords: Malignant neoplasms of independent (primary) multiple sites; Questionnaires; Surveys; Videos; Advanced Cancer
MeSH Terms: interventions — Surveys and Questionnaires; Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video 1: No EHR - Physician A (Experimental): Participant completes 5 questionnaires during an already-scheduled office visit.
  Participant then watches 2 short videos. After the first video, participant completes 3 questionnaires. After viewing the second video, participant completes 5 questionnaires.
  Interventions: Behavioral: Baseline Questionnaires; Other: Videos; Behavioral: Assessment Questionnaires
- Video 1: No EHR - Physician B (Experimental): Participant completes 5 questionnaires during an already-scheduled office visit.
  Participant then watches 2 short videos. After the first video, participant completes 3 questionnaires. After viewing the second video, participant completes 5 questionnaires.
  Interventions: Behavioral: Baseline Questionnaires; Other: Videos; Behavioral: Assessment Questionnaires
- Video 2: With EHR - Physician A (Experimental): Participant completes 5 questionnaires during an already-scheduled office visit.
  Participant then watches 2 short videos. After the first video, participant completes 3 questionnaires. After viewing the second video, participant completes 5 questionnaires.
  Interventions: Behavioral: Baseline Questionnaires; Other: Videos; Behavioral: Assessment Questionnaires
- Video 2: With EHR - Physician B (Experimental): Participant completes 5 questionnaires during an already-scheduled office visit.
  Participant then watches 2 short videos. After the first video, participant completes 3 questionnaires. After viewing the second video, participant completes 5 questionnaires.
  Interventions: Behavioral: Baseline Questionnaires; Other: Videos; Behavioral: Assessment Questionnaires

INTERVENTIONS:
Behavioral: Baseline Questionnaires — Participant completes 5 questionnaires during an already-scheduled office visit. Questionnaires ask about symptoms, physical and emotional health, and trust in the medical profession. These questionnaires should take about 17 minutes to complete.
  Other Names: Surveys
Other: Videos — Participant watches 2 short videos that show actors playing doctor and patient roles, discussing different cancer-related symptom treatment options. Each video is about 4 minutes long and discusses the same content, but setting of each video is different.
Behavioral: Assessment Questionnaires — After viewing first video, participant completes assessment questionnaire to evaluate their opinion of the physicians behavior. These questionnaires should take about 5 minutes to complete.
  After viewing second video, participant completes the same 3 assessment questionnaires. Participant also completes 2 additional questionnaires asking which physician participant would prefer as a primary physician and the satisfaction with health information technology use in their care.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn how patients feel about their doctors' attitudes toward supportive care and treatment options for advanced cancer patients.

DETAILED DESCRIPTION:
If you agree to take part in this study, during an already-scheduled office visit, you will complete 5 questionnaires about your symptoms, your physical and emotional health, and your trust in the medical profession. These questionnaires should take about 17 minutes to complete.

Study Groups:

After you have completed the first 5 questionnaires, you will be randomly assigned (as in the roll of the dice) to 1 of 4 groups.

Each group will watch 2 short videos that show actors playing doctor and patient roles, discussing different cancer-related symptom treatment options. Each video is about 4 minutes long and will discuss the same content, but setting of each video will be different.

After watching the first video, you will complete 3 questionnaires about your opinions of the doctor's behavior. These questionnaires should take about 5 minutes to complete.

After you watch the second video, you will complete the same 3 questionnaires. You will also complete 2 additional questionnaires about which doctor you would rather have as your doctor and why, and your opinion about the setting of the examination room in the video. It should take about 8 minutes to complete these questionnaires.

Length of Study:

It should take about 38 minutes to watch both videos and to complete all questionnaires. Your participation on this study will be over after you have completed the last questionnaire.

Other Information:

You must attend the study visit alone. Your family members should not be in the room with you while you are participating in the study. You may request to have family members remain in the room, but they must remain silent so that they do not influence your opinions.

This is an investigational study.

Up to 120 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of advanced cancer defined as locally advanced, recurrent or metastatic disease.
2. Outpatients (either new referrals or follow ups) seen in the Supportive Care Clinic.
3. Age >/= 18 years old
4. English speaking
5. Patients with normal cognitive status (Memorial Delirium Assessment Scale (MDAS) </=6/30) who are able to understand the nature and purpose of the study and have the ability to complete the consent process.

Exclusion Criteria:

1) Patients who are experiencing severe symptom distress, including severe emotional distress and cognitive dysfunction, which may interfere with study participation. This will be determined by the principle investigator and/or attending physician who is caring for the patient during that visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Participant's Rating of Physician's Compassion | 1 day
  Participant's rating of physician's compassion assessed by using a 5-item tool consisting of five 0-10 numerical rating scales assessing five dimensions: warm-cold, pleasant-unpleasant, compassionate distant, sensitive insensitive, caring-uncaring. The sum of the five scales gives a final score representing physician's compassion with a 0 to 50 scale.

SECONDARY OUTCOMES:
Participant's Rating of Physician Communication Skills | 1 day
  Participant's rating of physician communication skills assessed by using a 14-item tool consisting of 1 to 4 numerical rating scales assessing communication skills. The sum of these 14 scales gives a final score representing physician's communication skills with a 14 to 70 scale.
Participant's Rating of Physician's Professionalism | 1 day
  Participant's rating of physician's professionalism assessed by using a 4-item tool assessing politeness, listening, explaining the condition and treatment to the participant and participant's involvement in treatment decisions. Participant rates from poor to very good.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Haider, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org